CLINICAL TRIAL: NCT00298727
Title: Defining the Effect and Mediators of Two Knowledge Translation Strategies Designed to Alter Knowledge, Intent and Clinical Utilization of Rehabilitation Outcome Measures
Brief Title: The Effect and Mediators of Two Knowledge Translation Strategies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Joy MacDermid, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 152239
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Knowledge Transfer; Clinical Decision-making
Keywords: Knowledge transfer; Clinical decision-making; Outcome measures
MeSH Terms: interventions — Ships

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): SHIPS: Face-to-Face Workshop
  Interventions: Behavioral: SHIPS
- 2 (Active Comparator): ePBL: Online Problem-Based Course
  Interventions: Behavioral: ePBL

INTERVENTIONS:
Behavioral: SHIPS — Stakeholder-Hosted Interactive Problem-based Seminars
  Other Names: Face-to-Face workshop
  Arms: 1
Behavioral: ePBL — Online Problem-Based Course
  Arms: 2

SUMMARY:
Purpose: This study will compare the effectiveness and mediators of two different knowledge transfer (KT) interventions in terms of their impact on changing knowledge and behavior (utilization and clinical reasoning) related to health outcome measures.

DETAILED DESCRIPTION:
Interventions: Two different KT interventions with the same curriculum will be evaluated: 1. Stakeholder-Hosted Interactive Problem-Based Seminar (SHIPS), and 2. Online Problem-Based course (ePBL). SHIPs will consist of face-to-face PBL (Problem-based Learning) (2½ days) with outcome measure developers as facilitators, using 6 problems generated in consultation with participants. The ePBL will consist of a 6-week web-based course with 6 generic problems developed by content experts.

Outcome Measures: Baseline predictors including demographics, knowledge, attitudes/barriers regarding outcome measures and Readiness to Change will be assessed by self-report. Immediately post-intervention and 6 months later these will be re-administered. Primary qualitative and quantitative evaluations will be conducted 6-months post-intervention to assess the relative effectiveness of KT interventions and to identify elements that contribute to changing clinical behavior. Chart audits will determine the utilization of outcome measures (counts). Incorporation of outcome measures into clinical reasoning will be assessed using an innovative technique: chart-stimulated recall.

The Study Sample: Physical and Occupational Therapists (n=144; 80% power to detect an effect size of 0.5; alpha=0.05) will be recruited in partnership with the national professional associations.

Methods: SHIPS will be conducted in three urban centers in Canada. Participants will be block allocated by a minimization procedure to either of the two interventions to minimize any prognostic differences. Trained evaluators at each site will conduct chart audits and chart-stimulated recall. Trained interviewers will conduct semi-structured interviews focused on identifying critical elements in KT and implementing practice changes. Interviews will be transcribed verbatim.

Analyses: Analysis of covariance (ANCOVA), with baseline scores as a covariate, will be used to compare chart-stimulated recall scores at 6-months post-intervention. Secondary analyses will also use ANCOVA with the remaining potential predictors. Qualitative content analysis will be conducted iteratively until saturation is achieved.

Knowledge Impact and Transfer: A strategy for optimal transfer of health outcome measures into practice will be developed and shared with multiple disciplines involved in primary and specialty management of musculoskeletal and childhood disability. In addition, we will work with national professional organizations and Ministries of Health to use the knowledge from this study to support national initiatives on implementation and to assist with best KT practices in health service education.

ELIGIBILITY:
Inclusion Criteria:

* A valid license to practice physical or occupational therapy.
* Ability to communicate in English will be required.

Exclusion Criteria:

* Volunteers will be required to complete a knowledge pre-test in the format of a multiple-choice questionnaire. Those who are already knowledgeable, as determined by a score of 75% or greater, will be excluded to avoid ceiling effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Chart Audit Form (Utilization) | Up to 6 months post-intervention
Chart Stimulated Recall Data Collection Form | Up to 6 months post-intervention
Self-Efficacy Questionnaire | Up to 6 months post-intervention

SECONDARY OUTCOMES:
Readiness to Change Clinical Practice Scale | Up to 6 months post-intervention
Knowledge Test | Up to 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] MacDermid JC, Solomon P, Law M, Russell D, Stratford P. Defining the effect and mediators of two knowledge translation strategies designed to alter knowledge, intent and clinical utilization of rehabilitation outcome measures: a study protocol [NCT00298727]. Implement Sci. 2006 Jul 4;1:14. doi: 10.1186/1748-5908-1-14. PMID 16820055